CLINICAL TRIAL: NCT05025865
Title: Mechanisms by Which HA35 Regulates Muscle Protein Homeostasis in Healthy Controls
Brief Title: HA35 Acute Alcohol Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-486
Record Dates: First submitted 2021-08-18; First posted 2021-08-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Controls
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA35 Placebo Group (Placebo Comparator): 12 study participants will be given a placebo capsule to take once per day in the morning with breakfast for 3 days.
  Interventions: Drug: Placebo
- HA35 Treatment Group (Active Comparator): 12 study participants will be given an HA35 capsule to take once per day in the morning with breakfast for 3 days.
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Drug: Sodium Hyaluronate — Sodium Hyaluronate of molecular weight 35 kDa will be given in capsule form to the study participants.
  Other Names: HA35
  Arms: HA35 Treatment Group
Drug: Placebo — A placebo will be given in capsule form to study participants.
  Arms: HA35 Placebo Group

SUMMARY:
Eligible subjects will be asked to take a placebo/treatment capsule for a total of 3 days and then participate in a study visit on the fourth day. This study visit will include a medical exam, clinical labs, questionnaires, body composition measurements, and urine and stool collections. Additionally, participants will consume a sugar cocktail to measure their gut permeability, participate in an acute ethanol challenge, and undergo two muscle biopsies. The study will take approximately 3-4 hours and a designated driver will need to drive the participant home. On the fifth day, you will be asked to return to drop of the 24-hour urine collection.

DETAILED DESCRIPTION:
Interested subjects will be assessed for eligibility and a written informed consent will be obtained. The screening visit will consist of a medical exam, clinical labs (if not available in medical record), and questionnaires. Those who pass the screening will be eligible for a baseline visit (may be combined with screening if appropriate labs are already done). The baseline visit will include collection of blood, urine, and stool samples, body composition measurements, and randomization into either HA35 or placebo groups. Patients will be instructed to take the HA35 or placebo daily in the morning before breakfast 3 days prior to the day 4 visit. Patients will be informed that they will need to have a driver that is known to them for the day 4 visit. In the morning of the day 4 visit, confirmation of a driver will occur prior to starting study procedures. During the day 4 visit, patients will have an acute ethanol challenge where they will need to consume 2mL/kg of vodka in 100mL of juice in under 60 minutes. Muscle biopsies will be collected before and after the challenge and blood will be collected throughout the day. In addition, patients will be given lactulose/mannitol/sucralose/sucrose cocktail to measure gut permeability. The costs of any of these tests/procedures will not be billed to the patient and will be covered by the department. The participant will not be responsible for any costs.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol consumption of less than 7 drinks per week for women and less than 14 drinks per week for men
* Ability to understand and willingness to provide written consent

Exclusion Criteria:

* Any known chronic illness including but not limited to cancer (except non-melanoma skin cancer)
* Poorly controlled diabetes (Hemoglobin A1c >9.5 g/dl)
* Untreated hyper/hypothyroidism
* Uncontrolled hypertension or hypercholesterolemia
* End-stage renal disease
* Liver disease of any etiology
* Coronary artery disease or stroke
* Active intravenous drug use
* History of gastric bypass
* Medications known to alter muscle protein synthesis (systemic corticosteroids, tamoxifen, high dose estrogen, testosterone, or anabolic steroids)
* Pregnancy
* Past alcohol use disorder
* Abnormal clotting factors

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Aspartate Aminotransferase (AST) | Baseline to day 4
  change in units/liter (U/L)
Change in Alanine Aminotransferase (ALT) | Baseline to day 4
  change in units/liter (U/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided